CLINICAL TRIAL: NCT02697006
Title: Synchronized Cardiac Assist for Cardiogenic Shock. The SynCor Trial
Brief Title: Synchronized Cardiac Assist for Cardiogenic Shock
Status: Completed | Type: Observational
Sponsor: Xenios AG (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Organization: Fresenius Medical Care Deutschland GmbH (Industry)
Other Study IDs: Protocol 1.1 Version 1.0
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2020-09

CONDITIONS: Shock, Cardiogenic; High Risk Percutaneous Coronary Interventions
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: i-cor Synchronized Cardiac Assist Device — The i-cor Synchronized Cardiac Assist Device delivers pulsatile cardiac assist synchronized to the ECG during diastole and provides enhanced oxygenation through a membrane oxygenator.

SUMMARY:
The purpose of this study is to collect prospective safety and performance information for the i-COR® device using synchronized cardiac assist in the setting of combined heart-lung failure or in high risk percutaneous intervention procedures in catheterization lab.

ELIGIBILITY:
Inclusion Criteria:

Patients in cardiogenic shock in the setting of acute myocardial infarction

or

Patients undergoing high risk coronary revascularization procedures (e.g., multi-vessel disease, left main, or last patent conduit interventions) in the catheterization lab.

Cardiogenic shock is defined as

* Systolic blood pressure < 90 mmHg for at least 30 min or
* Inotropes are needed to maintain blood pressure > 90 mmHg or
* Clinical signs of heart insufficiency with pulmonary congestion or
* Signs of end organ hypoperfusion with at least one of the following criteria:
* Altered mental status
* cold, damp skin or extremities
* oliguria (≤ 30 mL/h)
* serum lactate > 2.0 mmol/L

Written consent of the patient or the legal caregiver

-

Exclusion Criteria:

* Age > 85 years
* Cardiac arrest out of hospital with return of spontaneous circulation (ROSC) > 10 min
* Coma with fixed pupils not induced by drugs;
* Mechanical causes for cardiogenic shock (ventricular septal defect of papillary muscle rupture)
* Non-cardiogenic causes of shock (bradycardia, sepsis, hypovolemia, etc.)
* Fever (Body temperature > 38.0 °C) or other evidence of sepsis
* Onset of cardiogenic shock > 6 h before enrollment;
* Lactate > 22 mmol/L;
* Massive pulmonary embolism;
* Severe peripheral arterial occlusive disease precluding insertion of femoral arterial or venous catheters
* Previous known aortic regurgitation greater than grade II
* Contra-indications for anticoagulation
* Severe hemolysis of any cause
* Patient is participating in an investigational drug or device study trial that has not reached the primary endpoint or that interferes with the current study endpoints.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiogenic shock or in high risk percutaneous intervention procedures in the cardiac catheterization lab
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04-30 (Actual); Study Completion 2019-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Liebetrau, Dr. med., Principal Investigator — Kerckhoff Klinik, Cardiology, Bad Nauheim, Germany
Locations (1):
- Kerckhoff Klinik, Bad Nauheim, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Risk PCI Group: Participants requiring ECG-synchronized cardiac assist in the setting of high-risk percutaneous intervention procedures in the catheterization lab
- Cardiogenic Shock: Participants requiring ECG-synchronized cardiac assist in the setting of combined heart-lung failure (cardiogenic shock)
Period: Overall Study
Arm/Group | High-Risk PCI Group | Cardiogenic Shock
Started | 34 | 13
Completed | 31 | 9
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Risk PCI Group | Cardiogenic Shock | Total
Number analyzed (Participants) | 34 | 13 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (10.9) | 67.5 (11.7) | 70.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 31 | 9 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 34 | 13 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device and Procedure Related Serious Adverse Events
Description: Acute safety defined as rates of device and procedure related serious adverse events up to 30 days post-intervention.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | High-Risk PCI Group | Cardiogenic Shock
Number analyzed (Participants) | 34 | 13
Participants | 11 | 5

2. Primary Outcome: Number of Participants Treated With Technical Success of the Device
Description: Technical success (defined as the ability to successfully deliver the i-COR® SYNCHRONIZED CARDIAC ASSIST device without serious adverse events).
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High-Risk PCI Group | Cardiogenic Shock
Number analyzed (Participants) | 34 | 13
Participants | 34 | 13

3. Primary Outcome: Number of Participants With Device Performance Success
Description: Device performance success (defined as the ability to establish synchronized pulsatile cardiac assist, enhance cardiac function and improve tissue oxygenation) assessed immediately post-procedure (acute) and serially as the device remains in place and provides cardiac support over time in each patient.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | High-Risk PCI Group | Cardiogenic Shock
Number analyzed (Participants) | 34 | 13
Participants | 34 | 13

ADVERSE EVENTS:
Time Frame: up to study exit at 30 days post-procedure, an average of 1 month
Arm/Group | High-Risk PCI Group | Cardiogenic Shock
All-Cause Mortality (participants affected / at risk) | 3/34 | 5/13
Serious Adverse Events (participants affected / at risk) | 10/34 | 5/13
Other Adverse Events (participants affected / at risk) | 0/34 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Risk PCI Group (N=34) | Cardiogenic Shock (N=13)
Bleeding event (Blood and lymphatic system disorders) | 8 (8) | 0 (0)
Wound infection groin (Infections and infestations) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deterioration in bispectral index (Nervous system disorders) | 1 (1) | 0 (0)
Death (Cardiac disorders) | 3 (3) | 5 (5)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0)
Syncope/Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Colonic impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower leg ischemia due to arterial clot (Vascular disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The low resistance puls kit oxygenator was not available at the inception of, nor the duration of the study, and therefore, efforts to demonstrate the physiological effect of ECG-synchronized, primarily diastolic assist cannot be determined by this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02697006/Prot_SAP_000.pdf